CLINICAL TRIAL: NCT00000866
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blind Trial to Evaluate the Safety and Immunogenicity of the Therion Recombinant Vaccinia-HIV-1 IIIB ENV/GAG/POL Vaccine (TCB-3B) and MN RGP 120/HIV-1 In Alum.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 014C; 10562 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Vaccinia Virus; Placebos; HIV-1; AIDS Vaccines; HIV Seronegativity; Genes, env; Genes, pol; Genes, gag; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections; Vaccinia

INTERVENTIONS:
Biological: MN rgp120/HIV-1
Biological: TBC-3B Vaccine

SUMMARY:
To evaluate the safety of administering Therion Recombinant Vaccinia-HIV-1 IIIB env/gag/pol Vaccine (TBC-3B) vaccinations to vaccinia-naive individuals. To evaluate the immunogenicity of priming with TBC-3B by the scarification, intradermal, and subcutaneous routes, followed by booster immunization of MN rgp120 HIV-1. To compare the immunogenicity of priming with TBC-3B in vaccinia-naive individuals to vaccinia-immune individuals.

In prior trials evaluating alternative methods of vaccine administration, scarification has been found to be an imprecise method of administration and allows only 1.0 - 2.5 microliters of immunogen to be given. Since it is not feasible to produce vaccine at concentrations higher than 10 to the 10th pfu/ml, this method limits the maximum deliverable dose. Intradermal and subcutaneous injection routes allow larger volumes of vaccinia to be given, i.e.: up to 200 microliters intradermally and up to 100 ml subcutaneously. In the present study, the initial priming dose will be the same administered by all 3 methods; however, the second priming dose administered at 2 months intradermally and subcutaneously will be 2 logs higher in order to achieve boosting of immune responses, particularly to gag and pol components of TBC-3B.

DETAILED DESCRIPTION:
In prior trials evaluating alternative methods of vaccine administration, scarification has been found to be an imprecise method of administration and allows only 1.0 - 2.5 microliters of immunogen to be given. Since it is not feasible to produce vaccine at concentrations higher than 10 to the 10th pfu/ml, this method limits the maximum deliverable dose. Intradermal and subcutaneous injection routes allow larger volumes of vaccinia to be given, i.e.: up to 200 microliters intradermally and up to 100 ml subcutaneously. In the present study, the initial priming dose will be the same administered by all 3 methods; however, the second priming dose administered at 2 months intradermally and subcutaneously will be 2 logs higher in order to achieve boosting of immune responses, particularly to gag and pol components of TBC-3B.

After volunteers are recruited, screened and enrolled in the study, they will be randomized to group C, D, or E. Each group will enroll 10 patients and 2 controls. The placebo control for TBC-3B will be standard vaccinia vaccination administered at doses no higher than that administered by scarification; the placebo control for MN rgp120 will be alum. Group C will receive undiluted TBC-3B by scarification, at months 0 and 2. Group D will receive diluted TBC-3B intradermally at month 0 and undiluted TBC-3B at month 2. Group E will receive diluted TBC-3B subcutaneously at month 0 and undiluted TBC-3B at month 2. At months 8 and 12 all groups will receive MN rgp 120/HIV-1 in alum intramuscularly.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Negative FDA-approved ELISA for HIV within 8 weeks of immunization.
* Normal history and physical examination.
* Negativity for Hepatitis B surface antigen.
* Availability for follow-up for planned duration of the study (18 months).

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Medical or psychiatric condition or occupational responsibilities that preclude subject compliance with the protocol. Specifically excluded are people with a history of suicide attempts, recent suicidal ideation or who have past or present psychosis.
* Active syphilis. NOTE: If the serology is documented to be a false positive or due to a remote (> 6 months) treated infection, the volunteer is eligible.
* Active tuberculosis. NOTE: Patients with a positive PPD and a normal chest X-ray showing no evidence of TB and not requiring INH therapy are eligible.
* Household contacts with, or occupational exposure to, people with any of the following:

Pregnancy. <12 months of age. Eczema or Immunodeficiency disease. Use of immunosuppressive medications.

Patients with the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, malignancy or autoimmune disease.
* History of cancer, unless there has been surgical excision followed by a sufficient observation period to give a reasonable assurance of cure.
* Any history of anaphylaxis or history of other serious adverse reactions to vaccines.
* History of serious allergic reaction to any substance, requiring hospitalization or emergent medical care (e.g., Stevens-Johnson syndrome, bronchospasm, or hypotension).
* Eczema within the past year.
* History of smallpox vaccination.
* Envelope bands on HIV-1 Western blot within 8 weeks of immunization.

Prior Medication: Excluded:

* Use of immunosuppressive.
* Live attenuated vaccines within 60 days of study.
* NOTE: Medically indicated subunit or killed vaccines (e.g. influenza, pneumococcal) do not exclude, but should be given at least 2 weeks prior to HIV immunizations.
* Experimental agents within 30 days prior to study.
* Prior receipt of HIV-1 vaccines or placebo recipient in a previous HIV vaccine trial.

Receipt of blood products or immunoglobulin within past 6 months.

Risk Behavior: Excluded:

* History of injection drug use within the last 12 months prior to enrollment.
* Higher or intermediate risk sexual behavior as defined by the AVEG.
* Lower risk sexual behavior as defined by AIDS Vaccine Evaluation Group (AVEG) procedures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36
Dates: Study Completion 1999-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Smith C, Study Chair
Locations (4):
- United States (4):
  - JHU AVEG, Baltimore, Maryland
  - St. Louis Univ. School of Medicine AVEG, St Louis, Missouri
  - Vanderbilt Univ. Hosp. AVEG, Nashville, Tennessee
  - UW - Seattle AVEG, Seattle, Washington

REFERENCES:
- [Background] Keefer MC, McElrath MJ, Weinhold K, Gorse GJ, Mulligan M, Francis D, Panicali D. A phase I trial of vaccina-eng/gag/pol (TBC-3B) given by alternative routes, boosted with rgp120. Int Conf AIDS. 1998;12:278 (abstract no 496/21199)